CLINICAL TRIAL: NCT04950660
Title: Oral Caffeine Decreases the Frequency of Opioid Demand in AIS Patients After Spinal Fusion
Brief Title: Oral Caffeine Use for Pain Management in AIS Patients After Spinal Fusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Anne Stuedemann, APRN III, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY00000775
Record Dates: First submitted 2021-06-15; First posted 2021-07-06 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, randomized control trial and will be double-blinded, with the patient, provider, and researcher blinded to the treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be a prospective, randomized control trial and will be double-blinded, with the patient, provider, and researcher blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caffeine arm (Active Comparator): Experimental Group: patient group (n = 34) receiving a 100 mg dose of caffeine (1/2 of a 200mg tablet to be taken whole or crushed), taken twice daily. This will be an adjuvant to their standard pain control.
  Interventions: Drug: Caffeine Tablet
- Placebo arm (Placebo Comparator): Control group: patient group (n = 34) receiving placebo compounded to look similar to the caffeine treatment, taken twice daily. This will be an adjuvant to their standard pain control.
  Interventions: Drug: Caffeine Tablet; Drug: Placebo

INTERVENTIONS:
Drug: Caffeine Tablet — Caffeine is approved by the FDA as a stimulant. A stimulant approved by the United States Food and Drug Administration (FDA) for the treatment to increase mental alertness and in combination with painkiller to treat migraine headaches. It is approved in the form of pill or tablet.
  Other Names: Caffeine
Drug: Placebo — Placebo, empty opaque dark blue blank capsule, taken twice daily. This will be an adjuvant to their standard pain control.
  Other Names: Blank
  Arms: Placebo arm

SUMMARY:
Prospective, randomized control trial To determine if oral caffeine decreases the frequency of opioid demand in children with adolescent idiopathic scoliosis after their spinal fusion surgery To compare pain scale ratings, number of requests for diazepam, average heart rate, average blood pressure, sex, age, ethnicity, post-op day of discharge, operative time, estimated intraoperative blood loss, remittance post-surgery, length of hospital stay, and segments fused during spinal fusion surgery.

DETAILED DESCRIPTION:
Because these receptors are so important for modifying pain and inflammation, caffeine has been added as an adjuvant to common analgesics, such as paracetamol, ibuprofen, and aspirin in the belief that it will enhance their analgesic efficacy. Most studies used paracetamol or ibuprofen with 100 mg to 130 mg caffeine, and the most common pain conditions studied were postoperative dental pain, postpartum pain, and headache. There was a small but statistically significant benefit with caffeine used at doses of 100 mg or more, which was not dependent on the pain condition or type of analgesic. Additionally, trials have shown superior efficacy of adding caffeine to ibuprofen instead of administering ibuprofen alone for treating acute pain, reflecting that caffeine is an effective analgesic adjuvant. The addition of caffeine (≥ 100 mg) to a standard dose of commonly used analgesics provides a small but important increase in the proportion of participants who experience a good level of pain relief.

Finally, the beneficial effects of caffeine on aerobic activity and resistance training performance are well documented. Studies have shown that caffeine ingestion resulted in significantly lower levels of soreness compared with placebo (p ≤ 0.05). A further beneficial effect of sustained caffeine ingestion in the days after the exercise bout is an attenuation of delayed onset muscle soreness. Orthopaedic surgery also causes muscle injury, and patients might benefit from caffeine's effect on lowering muscle soreness. Acute caffeine administration also has been shown to demonstrate increases in alertness, contentment, motivation to work, talkativeness, and energy. It also decreases muscle twitches. All of these effects would be beneficial in the post-operative period, especially for Adolescence Idiopathic Scoliosis (AIS) patients undergoing spinal fusion surgery in the orthopaedic department at Children's Mercy Hospital.

ELIGIBILITY:
Inclusion Criteria:

* must meet criteria for surgical correction of scoliosis
* must be able to swallow pills
* must have English as a primary language
* must possess mental capacity to understand purpose of the study
* patient must carry diagnosis of adolescent idiopathic scoliosis
* surgery must be performed via posterior approach
* operation performed by either Dr. John T. Anderson, Dr. Richard M. Schwend, Dr. Aaron Shaw, Dr. Michael Benvenuti
* post-surgical AIS patients from June 2019-June 2024
* the patient must be between the ages of 12 and 17 years old
* the patient and one of their biological parents or guardian(s) must give consent for patient to be included in this study
* Negative Suicide screen

Exclusion Criteria:

* obesity, as defined by a BMI at or above the 95th percentile
* weight below 40 kg
* any orthopedic diagnosis other than AIS
* revision spine surgery
* anterior or combined approach
* admission to PICU post-op
* use of Oxycodone post-op
* allergies to ibuprofen, caffeine, codeine, or diazepam
* history of renal disease
* history of a coagulation disorder
* history of cardiac dysrhythmia or open heart surgery
* history of Chronic Pain Syndrome or Complex Regional Pain Syndrome
* current use of oral central nervous system stimulant (e.g. methylphenidate)
* Positive Suicide screen

The following populations will be excluded:

* Children over the age of 18, or turning 18 during time of surgical treatment
* Children or parents unable to consent
* Individuals with cognitive delays
* Pregnant females
* Prisoners
* Wards of the state

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Stuedemann, APN, MSN, Principal Investigator — CHILDREN'S MERCY HOSPITALS & CLINICS
Locations (1):
- Children'S Mercy Hospitals & Clinic, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
only the research team will have access to study results. No IPD will be shared with anyone outside of the research team.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caffeine Arm | Placebo Arm
Started | 30 | 31
Completed | 24 | 27
Not Completed | 6 | 4
Not completed — Protocol Violation | 4 | 2
Not completed — Poor pain control, switch to Oxycodone | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Hypotension | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine Arm | Placebo Arm | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 27 | 51
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.25 (1.5) | 14.81 (1.4) | 14.55 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51
Weight [Mean (Standard Deviation); unit: Kg] — Population: Did not measure combined weight
  Kg | 53.8 (8.2) | 54.72 (7.1) | 54.29 (7.56)
Complications [Count of Participants; unit: Participants] | 0 | 0 | 0
Operative Time [Mean (Standard Deviation); unit: Minutes] | 230.92 (49.6) | 246.15 (43.4) | 238.98 (46.58)
Number of Segments Fused [Mean (Standard Deviation); unit: Number of segments] | 9.92 (2.1) | 10.52 (1.9) | 10.24 (1.98)

OUTCOME MEASURES:

1. Primary Outcome: Total Post Operative Oral Morphine Milligram Equivalents (MME)/Kilogram (Kg) for Hospital Stay
Description: Total Post Operative Oral Morphine milligram equivalents (MME)/kilogram (Kg) for Hospital Stay
Time Frame: For hospital stay up to 7 days
Measure: Mean (Standard Deviation); unit: MME/Kg
Groups:
- Caffeine Arm: Experimental Group: patient group (n = 24) receiving a 100 mg dose of caffeine (1/2 of a 200mg tablet to be taken whole or crushed), taken twice daily. This will be an adjuvant to their standard pain control.
  Caffeine Tablet: Caffeine is approved by the FDA as a stimulant. A stimulant approved by the United States Food and Drug Administration (FDA) for the treatment to increase mental alertness and in combination with painkiller to treat migraine headaches. It is approved in the form of pill or tablet.
- Placebo Arm: Control group: patient group (n = 27) receiving placebo compounded to look similar to the caffeine treatment, taken twice daily. This will be an adjuvant to their standard pain control.
  Caffeine Tablet: Caffeine is approved by the FDA as a stimulant. A stimulant approved by the United States Food and Drug Administration (FDA) for the treatment to increase mental alertness and in combination with painkiller to treat migraine headaches. It is approved in the form of pill or tablet.
  Placebo: Placebo, empty opaque dark blue blank capsule, taken twice daily. This will be an adjuvant to their standard pain control.
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
MME/Kg | 0.83 (0.41) | 0.92 (0.33)

2. Secondary Outcome: Mean Daily Verbal Analog Scale (VAS)
Description: Utilizing Verbal Analog Scale 0-10, 0 being no pain and 10 being severe pain
Time Frame: For hospital stay up to 7 days
Measure: Mean (Standard Deviation); unit: Units on a scale/day
Groups:
- Placebo Arm: Control group: patient group (n =27) receiving placebo compounded to look similar to the caffeine treatment, taken twice daily. This will be an adjuvant to their standard pain control.
  Caffeine Tablet: Caffeine is approved by the FDA as a stimulant. A stimulant approved by the United States Food and Drug Administration (FDA) for the treatment to increase mental alertness and in combination with painkiller to treat migraine headaches. It is approved in the form of pill or tablet.
  Placebo: Placebo, empty opaque dark blue blank capsule, taken twice daily. This will be an adjuvant to their standard pain control.
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
Units on a scale/day | 3.33 (1.65) | 3.51 (1.48)

3. Secondary Outcome: Average Heart Rate During Hospital Stay
Description: Documented heart rates which are then averaged over 24 hours
Time Frame: For hospital stay up to 7 days
Measure: Mean (Standard Deviation); unit: Beats per minute/day
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
Beats per minute/day | 78.8 (10.3) | 83.8 (12.4)

4. Secondary Outcome: Average Systolic Blood Pressure During Hospital Stay
Description: Documented systolic blood pressures which are then averaged over 24 hours
Time Frame: For hospital stay up to 7 days
Measure: Mean (Standard Deviation); unit: mmHg/day
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
mmHg/day | 98.3 (6.5) | 101.4 (6.6)

ADVERSE EVENTS:
Time Frame: 2-5 days postoperatively
Description: There were no documented complications, adverse events, or adverse drug reactions related to caffeine usage in this study.
Groups:
- Caffeine Arm: Experimental Group: patient group (n =24) receiving a 100 mg dose of caffeine (1/2 of a 200mg tablet to be taken whole or crushed), taken twice daily. This will be an adjuvant to their standard pain control.
  Caffeine Tablet: Caffeine is approved by the FDA as a stimulant. A stimulant approved by the United States Food and Drug Administration (FDA) for the treatment to increase mental alertness and in combination with painkiller to treat migraine headaches. It is approved in the form of pill or tablet.
Arm/Group | Caffeine Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04950660/Prot_SAP_000.pdf